CLINICAL TRIAL: NCT03676140
Title: A Cluster Randomised Trial of the Safety of Co-Administration of IDA (Ivermectin, Diethylcarbamazine and Albendazole) & Azithromycin for Integrated Treatment of Neglected Tropical Diseases
Brief Title: Safety of Co-administration of IDA and Azithromycin for NTDs ( ComboNTDs )
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lihir Medical Centre (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Oriol Mitja, Principal Investigator, Lihir Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ComboNTDs - CRT
Record Dates: First submitted 2018-09-16; First posted 2018-09-18 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Trachoma; Yaws; Lymphatic Filariases; Scabies; Strongyloidiasis
Keywords: Neglected Tropical Diseases
MeSH Terms: conditions — Trachoma; Yaws; Elephantiasis, Filarial; Scabies; Strongyloidiasis; Neglected Diseases | interventions — Albendazole; Ivermectin; Diethylcarbamazine; Azithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Separate Administration (Active Comparator): 'Albendazole on day 1' 'Ivermectin on day 1' 'Diethylcarbamazine on day 1' 'Azithromycin on day 8'
  Interventions: Drug: Albendazole on Day 1; Drug: Ivermectin on Day 1; Drug: Diethylcarbamazine on day 1; Drug: Azithromycin on Day 8
- Co-Administration (Experimental): 'Albendazole on day 1' 'Ivermectin on day 1' 'Diethylcarbamazine on day 1' 'Azithromycin on day 1'
  Interventions: Drug: Albendazole on Day 1; Drug: Ivermectin on Day 1; Drug: Diethylcarbamazine on day 1; Drug: Azithromycin on Day 1

INTERVENTIONS:
Drug: Albendazole on Day 1 — Albendazole 400 mg oral tablet Single Dose Treatment on D1
  Other Names: Albenza
Drug: Ivermectin on Day 1 — Ivermectin 200 µg/kg oral tablet Single Dose Treatment on Day 1
  Other Names: Mectizan
Drug: Diethylcarbamazine on day 1 — Diethylcarbamazine 6 mg/kg oral tablet Single Dose Treatment on Day 1
  Other Names: DEC-d1; Banocide
Drug: Azithromycin on Day 1 — Azithromycin 30mg/Kg oral tablet Single Dose Treatment On Day 1
  Other Names: Zithromax
  Arms: Co-Administration
Drug: Azithromycin on Day 8 — Azithromycin 30mg/Kg oral tablet Single Dose Treatment On Day 8
  Other Names: Zithromax
  Arms: Separate Administration

SUMMARY:
This is a cluster randomised trial evaluating the safety of co-administering Azithromycin alongside the new IDA (Ivermectin, Diethylcarbamazine, Albendazole) combination treatment for LF.

Treatment will be provided as a single dose Mass Drug Administration (MDA) to the whole community. Communities will be randomised to receive either treatment with IDA and Azithromycin on the same day or separately.

Active monitoring for adverse events will be conducted and the frequency of adverse events compared between individuals receiving combined MDA or separate MDA.

DETAILED DESCRIPTION:
Recent studies have shown that single-dose combination therapy with three antifilarial drugs (Ivermectin [IVE] + DEC + ALB) called IDA is superior to current regimens used in LF elimination and may help accelerate LF elimination. WHO guidelines have changed to recommend IDA in countries endemic for LF outside sub-Saharan Africa like Papua New Guinea.

Additional benefits of IVE are its activity against scabies and Strongyloides. Treatment with IVE has shown to reduce the high prevalence of scabies in a village and in randomized control trials elsewhere in the Pacific. Of particular importance was the finding that IVE was highly effective against Strongyloides with a >95% reduction in prevalence sustained for nine months.

Increasingly, the desirability of linking LF programs with other public health initiatives also based on MDA is being appreciated. The existing programmatic infrastructure developed for LF campaign presents an attractive vehicle for a demonstration project of integration of MDAs against multiple Neglected Tropical Diseases (NTDs). The macrolide antibiotic azithromycin (AZI) has been demonstrated to be highly effective as MDA for yaws control and AZI is a highly effective and well-tolerated antibiotic treatment for trachoma that is able to clear ocular infection with a single oral dose and is well tolerated.

Currently LF/STH/Scabies/strongyloides and yaws/trachoma are treated separately. Integration of these existing MDA programs has the potential to be highly cost-effective as a population health intervention. Integration includes both the safe co-administration of medicines and operational planning, and it is currently advocated by WHO.

ELIGIBILITY:
Inclusion Criteria:

* Able to give consent

Exclusion Criteria:

* Unable to give consent.
* Less than 5 years of age (not eligible for ivermectin)**
* Pregnant women (azithromycin only, not eligible for albendazole and ivermectin)
* Lactating women (Only administered azithromycin and albendazole, not eligible for ivermectin)**
* History of allergies to the drugs being studied
* Residents who cannot swallow tablets

Note that patients that are not eligible for a specific drug will receive all other treatments and will be followed up through the same procedure as the other participants drug therapy to try to track any AEs attributed to specific drug combinations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20000 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Self Reported Adverse Event | 7 Days
  The incidence of self-reported adverse events following MDA. We will collect data on the presence of common symptoms/signs prior to drug administration. All patients will be reviewed 24-48 hours after treatment and asked to report adverse events. We will calculate the proportion of newly occurring adverse events following treatment and calculate the whether the proportion of patients experiencing an adverse event differs between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy John, MD, Principal Investigator — National Department of Health of Papua New Guinea
Locations (1):
- Namatanai Hospital, Namatanai, Papua New Guinea

IPD SHARING:
Plan to Share IPD: No